CLINICAL TRIAL: NCT04867408
Title: EVEREST - IBD: Endoscopic Severity Image Recognition to Advance Research and Training in Inflammatory Bowel Disease
Brief Title: Endoscopic Severity Image Recognition to Advance Research and Training in Inflammatory Bowel Disease (EVEREST - IBD)
Status: Recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Wellcome/EPSRC Centre for Interventional and Surgical Sciences, University College London (Unknown)
Responsible Party: Sponsor
Other Study IDs: 299614
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Disease 1
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main group: Patients with/suspected Inflammatory Bowel Disease attending for an endoscopic procedure
- Control: Patients without Inflammatory Bowel disease attending for an endoscopic procedure

SUMMARY:
To develop and train a convolutional neural network to detect and characterize disease severity of inflammatory bowel disease during endoscopy

DETAILED DESCRIPTION:
To develop and train a Convolutional Neural Network to detect and characterize disease severity in inflammatory bowel disease during endoscopy. This initiative will inevitably establish a high-quality large image database. Our secondary study aims are therefore to use the images we collect to advance the field of deep learning and computer aided diagnosis in inflammatory bowel disease by establishing an image database. This will involve developing a framework combining deep learning and computer vision algorithms. The ultimate aim is to use the image database to produce high impact research outcomes and training resources leading to an improvement in the quality of endoscopy performed, reduce inter-observer variability in disease assessment and a reduction in missed bowel cancer rates and associated mortality.

ELIGIBILITY:
Inclusion Criteria:

* • Any adult patient aged 16 years or older who has consented to undergo endoscopic investigation where images are captured as part of routine clinical care.

Exclusion Criteria:

* • Any patient under the age of 16

  * Patients who are unable to give informed consent to undergo endoscopic investigation or those who do not wish their pseudo-anonymised images to be used

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inflammatory Bowel Disease (IBD) affects at least one in 250 people of the UK population and the prevalence is rising.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
To develop and train a convolutional neural network to detect and characterise disease severity of inflammatory bowel disease during endoscopy | 5 years
  To develop and train a convolutional neural network to detect and characterise disease severity of inflammatory bowel disease during endoscopy

SECONDARY OUTCOMES:
a) To explore whether Artificial Intelligence can predict response to IBD therapies | 5 years
  To explore whether Artificial Intelligence can predict response to IBD therapies
b) To develop an endoscopic image repository to advance training and standardisation in endoscopic detection and characterisation of IBD. | 5 years
  b) To develop an endoscopic image repository to advance training and standardisation
c) To develop and assess methodologies for training and quality assurance of IBD diagnostic endoscopy | 5 years
  To develop and assess methodologies for training and quality assurance of IBD
d) To evaluate comparisons in endoscopic image interpretation between endoscopist's | 5 years
  To evaluate comparisons in endoscopic image interpretation between endoscopist's
e) To develop deep learning algorithms and computer vision techniques to allow for automated measurement of quality metrics in endoscopy for IBD | 5 years
  To develop deep learning algorithms and computer vision techniques to allow for automated measurement of quality metrics in endoscopy for IBD
f) To create a future robust research platform to ensure the above objectives are continuously developed as novel imaging techniques emerge over time. | 5 years
  To create a future robust research platform to ensure the above objectives are continuously developed as novel imaging techniques emerge over time.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Sebastian, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull Royal Infirmary, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided